CLINICAL TRIAL: NCT02224963
Title: Improving Care Planning and Well-being in Older Adults With Macular Degeneration
Brief Title: Macular Degeneration and Aging Study
Acronym: MADAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Dartmouth-Hitchcock Medical Center (Other); Association for the Blind and Visually Impaired (Unknown)
Responsible Party: Principal Investigator, Silvia Sorensen, Research Associate Professor, University of Rochester
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: AG 032032
Record Dates: First submitted 2014-07-03; First posted 2014-08-25 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Age-related Macular Degeneration
Keywords: Aging,; Macular Degeneration,; Preparation for Future Care,; Psychological Well-being,; Problem Solving; Prevention; Mental Health Promotion
MeSH Terms: conditions — Macular Degeneration; Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Preventive Problem-Solving Training (Experimental): Preventive Problem-solving Training is an adaptation of Problem-Solving Therapy that builds problem-solving skills and then focuses these skills on potential future problems. It aims to reduce avoidance of contemplation of future needs and enhance gathering information, decision-making, and concrete planning about future needs.
  Interventions: Behavioral: Preventive Problem-Solving Training
- Life and Health Review (Active Comparator): Life and Health Review is an Enhanced Attention Control that provides classes and resource information modules, just as in intervention. It differs from the intervention in that we conduct an 8-session life and health review with subjects, in which they recount life experiences from childhood to the present.
  Interventions: Behavioral: Life and Health Review

INTERVENTIONS:
Behavioral: Preventive Problem-Solving Training — Preventive Problem-solving Training is an adaptation of Problem-Solving Therapy that builds problem-solving skills and then focuses these skills on potential future problems. It aims to reduce avoidance of contemplation of future needs and enhance gathering information, decision-making, and concrete planning about future needs.
  Arms: Preventive Problem-Solving Training
Behavioral: Life and Health Review — Life and Health Review is an Enhanced Attention Control that provides classes and resource information modules, just as in intervention. It differs from the intervention in that we conduct an 8-session life and health review with subjects, in which they recount life experiences from childhood to the present.
  Arms: Life and Health Review

SUMMARY:
The purpose of this randomized trial is to examine the effectiveness of a psycho-social "Preventive Problem Solving Intervention" on emotional well-being, change in future outlook, and vision functioning in 250 Age-related Macular Degeneration patients 60 and older.

DETAILED DESCRIPTION:
Loss of independence and valued activities places Age-related Macular Degeneration (AMD) patients at increased risk for depression, anxiety, and disability. Patients' emotional and behavioral responses to AMD can exacerbate the long-term health threat of the disease and contribute to preventable health care costs, loss of productivity, and burden to family members.This is a randomized controlled trial of a psycho-social intervention that addresses three mental health promotion goals: (1) increase emotional well-being, (2) improve future outlook, and (3) protect or enhance current and future-oriented functioning.

The trial examines the effects of the PREPSI for 250 AMD patients, 60 and older, regardless of actual vision acuity. All study participants receive 4 group-based vision education classes and resource information. Subjects are then randomized to Preventive Problem Solving Intervention (PREPSI) consisting of 8 sessions with certified problem-solving trainers or to an Enhanced Attention Control arm.

Assessors blind to treatment condition measure Psychological Well-being immediately post-intervention (Week 16) and at 6-month follow-up, Change in Future Outlook, including Preparation for Future Care from baseline to 16 week and 6-month follow-up, and Vision Functioning at 6 month follow-up. Measures include the Psychological Well-being Scale (Ryff & Keyes, 1995), the Preparation of Future Care Needs Scale (Sörensen & Pinquart, 2001), and the National Eye Institute Vision Functioning Questionnaire-25 (Stelmack, Stelmack, & Massof, 2002). The primary hypothesis is that PREPSI participants will report greater Psychological Well-being and more Preparation for Future Care immediately post-intervention (at 16 weeks) and at 6-month follow-up.

The PREPSI is a short, standardized modification of problem-solving therapy that trains participants to identify and clearly define current and future problems, and then generate, evaluate, choose, and implement solutions. The long-term goal of the investigators research program is to improve quality of life in late adulthood by conducting basic and translational research on preventive future planning.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AMD
* 60 years and older
* Able to communicate in English.

Exclusion Criteria:

* Significant cognitive impairment at baseline (total score on Mini Mental State Exam (MMSE) for the Blind <18, equivalent to <21 in the regular MMSE);
* Residence in a nursing home (assisted living facilities are acceptable);
* Patient is acutely suicidal or psychotic

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2009-05 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Psychological Well-being | at 16 weeks (immediately post-intervention)
  The 42-item multidimensional Psychological Well-Being scale (PWB) will assess 6 dimensions of PWB: Autonomy, Environmental Mastery, Personal Growth, Positive Relations With Others, Purpose In Life, and Self-Acceptance. The PWB is a Likert-scored self-report measure, with anchors of "1-disagree strongly" and "6-agree strongly."
Psychological Well-being | at 6-month follow-up
  The 42-item multidimensional Psychological Well-Being scale (PWB) will assess 6 dimensions of PWB: Autonomy, Environmental Mastery, Personal Growth, Positive Relations With Others, Purpose In Life, and Self-Acceptance. The PWB is a Likert-scored self-report measure, with anchors of "1-disagree strongly" and "6-agree strongly."

SECONDARY OUTCOMES:
Change in Preparation for Future Care | from baseline to 16 weeks (immediately post-intervention)
  Preparation for Future Care Measure (PFCM) consists of 29 items in five subscales that assess specific behaviors representative of each of five processes observed in PFC: Awareness of care needs, Gathering Information, Deciding on Preferences, Making Concrete Plans, and Avoidance. It is rated on a fiv-point Likert Scale
Preparation for Future Care | at 6-month follow-up
  Preparation for Future Care Measure (PFCM) consists of 29 items in five subscales that assess specific behaviors representative of each of five processes observed in PFC: Awareness of care needs, Gathering Information, Deciding on Preferences, Making Concrete Plans, and Avoidance. It is rated on a fiv-point Likert Scale

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Sörensen, PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States